CLINICAL TRIAL: NCT03816215
Title: Volunteering as an Intervention to Reduce Depression Among Adolescents: Investigating Neurobiological Mechanisms
Brief Title: Volunteering as an Intervention to Reduce Depression Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00053435
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2020-03

CONDITIONS: Depression; Adolescent Behavior; Depressive Symptoms
Keywords: Adolescents; FMRI; volunteerism
MeSH Terms: conditions — Depression; Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescent Participants (Experimental): Participants will be assigned to participate in community service (from a menu of options) for 30 hours.
  Interventions: Behavioral: Volunteer experience

INTERVENTIONS:
Behavioral: Volunteer experience — Participants will be assigned to a meaningful volunteer experience from a menu of local options (e.g., volunteering at an animal shelter or in a library) for 30 hours.

SUMMARY:
The purpose of the present study is to test in a preliminary manner an innovative strategy for treating depression among adolescents (alongside existing therapy) using community volunteerism.

DETAILED DESCRIPTION:
The purpose of the present study is to test in a preliminary manner an innovative strategy for treating depression among adolescents (alongside existing therapy) using community volunteerism. In addition, this study will test a potential mechanism by which volunteering might decrease depressive symptoms: increasing psychosocial assets, specifically decreasing self-orientation and increasing an orientation toward others. This will be measured through self-report as well as using functional magnetic resonance imaging (fMRI). This study will be the first study to explore how neural response patterns are potentially altered by intense experiences with volunteerism among depressed adolescents.

ELIGIBILITY:
Inclusion Criteria:

* age 14-20
* new mild to moderate depression diagnosis (single episode)
* new mild to moderate anxiety diagnosis
* new adjustment disorder diagnosis
* have been in treatment for < 8 months
* right-handed

Exclusion Criteria:

* history of recurrent depressive, anxiety or adjustment disorder episodes
* have been in treatment > 8 months
* left-handed
* expressing suicidal ideation
* claustrophobia
* any contraindications for completing an MRI scan

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Participant recruitment | 6 months
  Number of participants screened (reported by clinical mental health providers)
Participant retention | 6 months
  Number of participants retained in full study
Depressive symptoms (Beck Depression Inventory) | 6 months
  Beck Depression Inventory to measure depressive symptoms. Each item is rated on a 4-point scale ranging from 0 to 3. The minimum total score is 0 and the maximum total score is 63. Higher scores denote worse outcome

SECONDARY OUTCOMES:
Strength of Connectivity in DMN (Default Mode Network) | 6 months
  Default Mode Network Connectivity will be measured using fMRI at rest and while processing emotional pictures before and after volunteering intervention. The strength of connectivity within the DMN will be calculated by averaging attributes for each node in the DMN.
Hope scale (Abler et al., 2017) | 6 months
  Hope scale (Abler et al., 2017) will be measured on a scale from 1 (strongly disagree) to 5 (strongly agree). Items will be averaged; higher scores denote better outcome (more hope).
Beck Hopelessness Inventory | 6 months
  Beck Hopelessness Inventory will be used (scored from 1-20; higher score denotes worse outcome).
Self-efficacy | 6 months
  NIH toolbox measure from 1 (never) to 5 (very often); scores will be averaged and high score indicates more self-efficacy.
Orientation Toward Others | 6 months
  5 point scale from 1=strongly disagree to 5=strongly agree. Scores will be averaged; higher score denotes more orientation toward others.
Empathy | 6 months
  IRI (Interpersonal Reactivity Index) subscale to measure empathy on a 5 point scale from 1- strongly disagree to 5 -strongly agree. Scores will be averaged; higher score denotes more empathy.

OTHER OUTCOMES:
Experience in Volunteering | 6 months
  Measured through the Inventory of Service Experience (Taylor & Pancer, 2007) on a scale from 1 (strongly disagree) to 5 (strongly agree). Scores will be averaged for subscales of the measure. Higher score denotes better outcomes (more positive experiences with volunteering).

CONTACTS AND LOCATIONS:
Overall Officials: Parissa Ballard, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Trinity Center, Inc, Winston-Salem, North Carolina
  - TriCare, PA, Winston-Salem, North Carolina
  - Private practice, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beck, J. S. (2011). Cognitive behavior therapy: Basics and beyond: Guilford Press
- [Background] Beesdo K, Hofler M, Leibenluft E, Lieb R, Bauer M, Pfennig A. Mood episodes and mood disorders: patterns of incidence and conversion in the first three decades of life. Bipolar Disord. 2009 Sep;11(6):637-49. doi: 10.1111/j.1399-5618.2009.00738.x. PMID 19689506
- [Background] Butler AC, Chapman JE, Forman EM, Beck AT. The empirical status of cognitive-behavioral therapy: a review of meta-analyses. Clin Psychol Rev. 2006 Jan;26(1):17-31. doi: 10.1016/j.cpr.2005.07.003. Epub 2005 Sep 30. PMID 16199119
- [Background] Gudayol-Ferre E, Pero-Cebollero M, Gonzalez-Garrido AA, Guardia-Olmos J. Changes in brain connectivity related to the treatment of depression measured through fMRI: a systematic review. Front Hum Neurosci. 2015 Nov 3;9:582. doi: 10.3389/fnhum.2015.00582. eCollection 2015. PMID 26578927
- [Background] Kessler RC, Avenevoli S, Ries Merikangas K. Mood disorders in children and adolescents: an epidemiologic perspective. Biol Psychiatry. 2001 Jun 15;49(12):1002-14. doi: 10.1016/s0006-3223(01)01129-5. PMID 11430842
- [Background] Sheline YI, Barch DM, Price JL, Rundle MM, Vaishnavi SN, Snyder AZ, Mintun MA, Wang S, Coalson RS, Raichle ME. The default mode network and self-referential processes in depression. Proc Natl Acad Sci U S A. 2009 Feb 10;106(6):1942-7. doi: 10.1073/pnas.0812686106. Epub 2009 Jan 26. PMID 19171889

DOCUMENTS (1):
  • Informed Consent Form (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT03816215/ICF_000.pdf